CLINICAL TRIAL: NCT00857571
Title: An Open-Label Randomized Incomplete Block Four-Way Crossover Study To Evaluate The Dose Response Of PF-02413873 Tablets And PF-02413873 Suspension.
Brief Title: A Four-Way Cross-Over Study To Compare The Plasma Concentrations Of PF-02413873 After Oral Administration Of Several Doses As Suspension And As Tablets.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B0461003
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Healthy
Keywords: Dose Response Bioavailability Study
MeSH Terms: interventions — Suspensions; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Suspension (Experimental): PF-02413873 suspension
  Interventions: Drug: 150 mg Suspension; Drug: 30 mg Suspension; Drug: 400 mg Suspension; Drug: 5 mg Suspension; Drug: 750 mg Suspension
- Tablet (Experimental): PF-02413873 Phase 2 Tablets
  Interventions: Drug: 150 mg Tablet; Drug: 30 mg Tablet; Drug: 400 mg Tablet; Drug: 5 mg Tablet; Drug: 750 mg Tablet

INTERVENTIONS:
Drug: 150 mg Suspension — Single oral dose of 150 mg of PF-02413873 suspension
  Arms: Suspension
Drug: 30 mg Suspension — Single oral dose of 30 mg of PF-02413873 suspension
  Arms: Suspension
Drug: 400 mg Suspension — Single oral dose of 400 mg of PF-02413873 suspension
  Arms: Suspension
Drug: 5 mg Suspension — Single oral dose of 5 mg of PF-02413873 suspension
  Arms: Suspension
Drug: 750 mg Suspension — Single oral dose of 750 mg of PF-02413873 suspension
  Arms: Suspension
Drug: 150 mg Tablet — Single oral dose of 150 mg of PF-02413873 tablets
  Arms: Tablet
Drug: 30 mg Tablet — Single oral dose of 30 mg of PF-02413873 tablets
  Arms: Tablet
Drug: 400 mg Tablet — Single oral dose of 400 mg of PF-02413873 tablets
  Arms: Tablet
Drug: 5 mg Tablet — Single oral dose of 5 mg of PF-02413873 tablets
  Arms: Tablet
Drug: 750 mg Tablet — Single oral dose of 750 mg of PF-02413873 tablets
  Arms: Tablet

SUMMARY:
The study compares the plasma concentrations of PF-02413873 after administration of several doses as suspension and as tablets

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers.
* Female volunteers have to be of non-childbearing potential

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Cmax, AUCinf | June - July 2009

SECONDARY OUTCOMES:
Tmax, Tlag, AUClast, AUCt, t½, Frel. | June-July 2009

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0461003